CLINICAL TRIAL: NCT06403917
Title: Evaluation of Breast Cancer Screening Program in Assiut Governorate "Egyptian Women Health Initiative"
Brief Title: Evaluation of Breast Cancer Screening Program at Assiut Governorate
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Essa, dr halaa saad essa, Assiut University
Other Study IDs: Evaluation of BC program
Record Dates: First submitted 2024-04-27; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of breast screening — Evaluation of breast screening program at egyptian women health intiaive

SUMMARY:
1. To evaluate the ability of breast clinical examination as screening tool to detect early and advanced stages of breast cancer.
2. To determine the percentage of breast cancer confirmed cases among women screened at women health campaign in Assiut governorate.
3. To determine drop out from referral system among screening program.
4. Identify the healthcare providers knowledge about breast cancer and screening tools, perception, practice and barriers in delivering the program

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed cancer and the leading cause of cancer death in females worldwide, Despite major efforts at early detection and new treatments, breast cancer claims the lives of over 520,000 women every year [1] with an estimated 2.3 million new cancer cases (1 in 4 new cancer cases) and 685,000 cancer deaths (1 in 6 deaths) in 2020.

Breast cancer incidence rates varied by nearly 4-fold across WHO areas. The highest incidence rates (per 100,000) were found in Australia/New Zealand (95.5), Western Europe (90.7), and Northern America (89.4), while the lowest rates were in South-Central Asia (26.2), Middle and Eastern Africa (33), and Central America (39.5). In contrast, the highest breast cancer mortality rates were recorded in Melanesia (37.5), Polynesia and Western Africa (22.3), and the Caribbean (18.9), while the lowest rates were found in Eastern Asia (9.8), Central America (10.4), and Australia/New Zealand standardized breast cancer incidence rate (per 100,000) increased from 106 (1975) to 142 (1999), decreased to 128 (2004), and then slowly increased to 137 (per 100,000) in 2019. Similar broad temporal trend patterns were observed in other western countries.[2] Incidence rates are rising in South America, Africa, and Asia where rates were historically low. Worldwide, an estimated 2,964,197 new female breast cancer cases are projected to occur in 2040, a 31% increase from the corresponding 2,260,127 cases in 2020. [3,4] Breast Cancer in Arab Countries From available data from the years 2010, 2013, and most recently 2020, breast cancer is thought to be the most common malignancy diagnosed in Arab women, estimating somewhere between 14-42% of all tumors [5 ,6]in some reports, and between 17.7-19% of all new cancers in others [7] depending on individual countries and type of reports reviewed.

In Egypt In Egypt, breast cancer is the most common malignancy in women, accounting for 38.8% of cancers in this population, with the estimated number of breast cancer cases nearly 22,700 in 2020 and forecasted to be approximately 46,000 in 2050. It is estimated that the breast cancer mortality rate is around 11%, being the second cause of cancer-related mortality after liver cancer.[9] Early diagnosis (in symptomatic populations) and screening (in asymptomatic populations) are the two main components of cancer early-detection programs, as defined by the WHO, to reduce the incidence of advanced cancer and mortality. In low- and middle-income countries, where cancer is diagnosed in advanced stages and allocated resources are limited, it is highly recommended that cancer control programs include the following elements: [1] targeted outreach/education promotion and [2] efforts to encourage clinical breast examination for at-risk groups, with or without opportunistic mammographic screening. This is to keep with the goal of downsizing symptomatic disease and/or asymptomatic disease in high-risk groups.[10] Breast self-examination (BSE), clinical breast examination (CBE) by a physician, and mammography are three instruments recommended for breast cancer screening. BSE is highly useful in breast cancer screening as it is cheap, easy, confidential, uncomplicated, and without the need for special equipment [11] Clinical Breast Examination (CBE) is defined as the examination of a woman's breasts by a healthcare professional, such as a breast surgeon, family physician or breast care nurse who is trained to recognize many different types of abnormalities and warning signs in the breast [12] Screening mammography is a low-dose X-ray examination of a woman's breasts used to detect BC when that cancer is too small to be felt as a lump. Screening mammography is very useful as it reduces mortality from BC by about 20%-35% in women aged 50-69 years and slightly less in women aged 40-49 years at a period of 14 years of follow-up [10].

In Egypt, facilities for mammographic screening are available in the major governmental and private hospitals and delivered through mobile units equipped with digital mammography units. Despite these mobile units, which increase the presence in rural areas and less affluent areas, barriers to accessing mammography still exist [13].

Delays to breast cancer treatment of greater than three months have been associated with more advanced disease stage at diagnosis and poorer survival. At the same time, education of primary care providers to recognize the early signs and symptoms of breast cancer is necessary for prompt referral through the healthcare system [14].

A retrospective analysis of cancer screening data from 2012 to 2019 was carried out in Jeddah, Saudi Arabia Of the 16000 women invited from 2012 to 2019, a total of 1911 (11.9%) participated. The majority of women (68.8%) were between 40 and 55 years old. Based on the screening process results, 26.6%, 40.1%, 9.7%, 1.3%, 0.7%, and 5.2% of women had BI-RADS scores of R1, R2, R3, R4, R5, and R0 respectively The remaining 16.3% did not have mammogram records. The recall rate, or the percentage of women who underwent further evaluation, was 19.9%; 18.9% underwent a biopsy procedure. In addition, 1.6% of women had cancer screen-detected, although only 0.7% were diagnosed with breast cancer.[15] A case-control study to evaluate the impact of the breast screening program on mortality in England. The study dataset had a total of 9550 cases and 17,993 controls; the main objective was to evaluate the effect of mammography screening on breast cancer mortality. This study showed that the breast screening programs in England continues to play an important role in the control of breast cancer. The effect of screening within the NHS BSP in England is stronger and longer lasting in women aged 65 or over, but it remains highly relevant for younger women. [16] In Egypt, the first national screening program, the Women Health Outreach Program, was initiated in October 2007. It was a government-funded program that offered free mammograms for Egyptian women aged > 45 and screening for diabetes, hypertension, and obesity. This was approached using mammography vans, equipped with a full-field digital mammography machine, and a dedicated computer system linked to the National Breast Screening Center. Free treatment was offered for cases in which breast cancer was detected. From October 2007 to February 2009, 20,098 women in three governorates were screened for breast cancer.[13][17] (Egypt is divided into 27 governorates, the highest tier of the country's jurisdiction hierarchy.) With the launch of the 100 Million Healthy Lives national initiative, more efforts were directed to control breast cancer in Egypt. In July 2019, a nationwide campaign was started in 9 governorates (Alexandria, Port Said, Matrouh, Qalyubia, Beheira, Assiut, Fayoum, South Sinai, and Damietta) and extended after 2 months to another 11 governorates (Cairo, North Sinai, the Red Sea, Ismailia, Suez, Kafr El-Sheikh, Menoufia, Beni Suef, Sohag, Luxor, and Aswan), and then after 2 more months, to the remaining 7 governorates (Giza, the New Valley, Gharbia, Dakahlia, Sharqia, Minya, and Qena). The main objectives of this campaign are to promote breast cancer awareness and the importance of early diagnosis, screening for breast cancer and treatment of diagnosed cases according to recent protocols. Suspected cases are referred for further investigation and treatment at no cost for the participants. The media center for the Council of Ministers announced that 8.5 million women had been examined by October 20, 2020, from all over Egypt, with the aim of reaching 31 million women. [18]

ELIGIBILITY:
Inclusion Criteria:A multi-stage stratified random sampling technique will be used to select the sample. Sites providing breast cancer screening service at Assiut governorate will be classified into primary health care unit and secondary hospitals.

Primary health care units providing breast cancer screening service at Assiut governorate will be stratified in to rural, urban units. Two rural and two urban units will be randomly selected. Women at each unit will be classified according to age into below 38 years and above 38 years. A proportionate sample will be taken from each group.

-

Exclusion Criteria:age below 18 year.

-

Ages: 18 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — females above18
Study Population: women coming to breast screening program at assiut governorate
Sampling Method: Probability Sample
Enrollment: 15000000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
1-To evaluate the ability of breast clinical examination as screening tool to detect early and advanced stages of breast cancer. | one year
  1. Retention rate The estimated percentage of women above18 y who returned for screening within 12months %
  2. Annual screening rate:The estimated percentage % of women above18 y who returned to screen within 18 months of their previous screen.

SECONDARY OUTCOMES:
2-To determine the percentage of breast cancer confirmed cases among women screened at women health campaign in Assiut governorate | one year
  1. Invasive cancer detection rate Number of invasive cancers detected per 1,000 screens.
  Non-malignant biopsy rate Number of non-malignant open and core biopsies per 1,000 screens (b) Percentage of non-malignant biopsies which were open surgical biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Faten Rabie, PHD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forouzanfar MH, Foreman KJ, Delossantos AM, Lozano R, Lopez AD, Murray CJ, Naghavi M. Breast and cervical cancer in 187 countries between 1980 and 2010: a systematic analysis. Lancet. 2011 Oct 22;378(9801):1461-84. doi: 10.1016/S0140-6736(11)61351-2. Epub 2011 Sep 14. PMID 21924486